CLINICAL TRIAL: NCT00849810
Title: Comparative Effects of Nebivolol Versus Metoprolol on 24-hour Blood Pressures and Basal Metabolic Rate: An Open-Label Study
Brief Title: Comparing the Effects of Two Beta Blockers,Metoprolol and Nebivolol,on Ambulatory Blood Pressure and Basal Metabolic Rate
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty with recruiting willing participants.
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Deborah Minor, Professor of Medicine, University of Mississippi Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0002
Record Dates: First submitted 2009-02-02; First posted 2009-02-24 (Estimated); Results first posted 2013-03-19 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Hypertension
Keywords: Hypertension; Beta-blockers; Ambulatory blood pressure; Basal metabolic rate; Quality of life
MeSH Terms: conditions — Hypertension | interventions — Metoprolol; Nebivolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metoprolol to nebivolol (Experimental): metoprolol 25-200mg at a stable daily dose for 4 weeks, then change to nebivolol at a comparable stable dose (5-20 mg) for 4 -5 weeks.
  Interventions: Drug: Metoprolol; Drug: Nebivolol

INTERVENTIONS:
Drug: Metoprolol — Metoprolol tablets 25-200 mg daily times four weeks. Nebivolol daily for 4-5 weeks
  Other Names: Nebivolol is bystolic; Metoprolol is lopressor
Drug: Nebivolol — 5 - 20 mg daily, at a stable dose for 4 to 5 weeks

SUMMARY:
The purpose of the study is to compare the effects of nebivolol and metoprolol on 24-hour ambulatory blood pressure characteristics and basal metabolic rates in patients with hypertension.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* currently be treated at a University of MS Medical Center Internal Medicine Clinics
* currently taking metoprolol succinate for hypertension
* have their hypertension controlled (<140/90).

Exclusion Criteria:

* uncontrolled hypertension
* severe renal or moderate hepatic impairment
* currently taking CYP 2D6 inducers/inhibitors
* recent stroke (less than 6 months)
* recent myocardial infarction (less than 6 months)
* congestive heart failure
* diagnosed obstructive sleep apnea
* atrial fibrillation
* arm circumference >50 cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Minor, PharmD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 11/2008-4/2009, 472 patient were prescribed metoprolol succinate. During screening, metoprolol succinate was discontinued in 87 patients and 177 were excluded (obstacles to visits, competency issues). A national shortage of metoprolol succinate caused discontinuation in mant patients. One patient was enrolled and completed the study.
Groups:
- Metoprolol to Nebivolol: Patients entered the study on metoprolol succinate, at stable dose of dose of 25-200mg daily for 4 weeks. Patients had ambulatory blood pressure assessment at their current dose and then were changed to a comparable dose of nebivolol. Ambulatory blood pressure assessment was repeated after approximately 4 to 5 weeks, at a stable dose.
  Metoprolol : Metoprolol tablets 25-200 mg daily times four weeks. Nebivolol daily for 4-5 weeks, 5-20 mg.
Period: Overall Study
Arm/Group | Metoprolol to Nebivolol
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Metoprolol to Nebivolol
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome is Pre- and Post-treatment Ambulatory Blood Pressure.
Time Frame: 4 weeks (pre- and post-treatment)
Measure: Mean (Standard Deviation); unit: mm HG
Arm/Group | Metoprolol to Nebivolol
Number analyzed (Participants) | 1
mm HG
  SBP ABPM on metoprolol | 122
  DBP ABPM on metoprolol | 72
  SBP ABPM on nebivolol | 122
  DBP ABPM on nebivolol | 71

ADVERSE EVENTS:
Arm/Group | Metoprolol to Nebivolol
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No